CLINICAL TRIAL: NCT03674944
Title: Targeting Emotional Eating and Weight Loss in Adolescents
Brief Title: FRESH-TEEN: Families Responsibility Education Support Health for Teens
Acronym: FRESH-TEEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Minnesota (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kerri Boutelle, Kerri Boutelle, Ph.D., Professor, Departments of Pediatrics and Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 180417; R01DK116616 (NIH)
Record Dates: First submitted 2018-08-22; First posted 2018-09-18 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Overeating; Treatment; Body Mass Index; Intervention; Behavioral Treatment; Dialectical Behavior Therapy; Emotion Regulation
MeSH Terms: conditions — Overweight; Obesity; Hyperphagia; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Weight Loss (BWL) + Emotion Regulation (ER) (Experimental): This program includes: 1) Dialectical Behavior Therapy (DBT) skills 2) Behavioral coaching 3) Emotional Focused Parent Training (EFPT) 4) Behavioral Weight Loss (BWL) skills.
  Interventions: Behavioral: Behavioral Weight Loss (BWL) + Emotion Regulation (ER); Behavioral: Behavioral Weight Loss (BWL)
- Behavioral Weight Loss (BWL) (Active Comparator): This program includes information about diet and physical activity education, in addition to parent management skills, and behavioral modification principles including: modeling, reinforcement, and operant conditioning.
  Interventions: Behavioral: Behavioral Weight Loss (BWL)

INTERVENTIONS:
Behavioral: Behavioral Weight Loss (BWL) + Emotion Regulation (ER) — The BWL + ER program will teach Dialectical Behavior Therapy (DBT) skills (dialectical abstinence, emotion regulation skills, mindfulness, and distress tolerance) to the adolescent and parent group sessions. Parents are expected to model skill usage and DBT language with their teen to reinforce the skills at home. Adolescents and parents will track emotions and DBT skills used in diary cards which will be provided. Emotion-Focused Parent Training (EFPT) will be provided to the parents at each session to train the parent to support the adolescent in processing emotions, increasing parental emotion self-efficacy, promoting positive parent-adolescent relationships, and reducing the need for dysfunctional emotion regulation behaviors.Behavior coaching will be provided to the adolescent and parent to encourage compliance and review skills after each session (DBT or BWL).
  Arms: Behavioral Weight Loss (BWL) + Emotion Regulation (ER)
Behavioral: Behavioral Weight Loss (BWL) — All participants will be instructed to consume an energy restricted diet based on initial body weight. Participants will be instructed to record and self-monitor their food intake. The physical activity component will focus on increasing both lifestyle activity and structured exercise programs. Behavior change recommendations will include: self-monitoring, goal setting, managing high-risk situations, and relapse prevention. Parenting skills will be discussed during parent group sessions which will encourage parents to adopt authoritative parenting styles with regard to eating and exercise behaviors. Parents will also learn about behavioral modification principles, including modeling, reinforcement, and operant conditioning. Behavior coaching will be provided to the adolescent and parent after each session to encourage compliance, discuss completed homework, review habit books to praise efforts and give feedback for areas of improvement.
  Other Names: BWL

SUMMARY:
The objective of this proposed study is to collect initial efficacy data on a behavioral weight loss (BWL) program for teens, which also includes emotion regulation strategies (ER), to standard BWL.

DETAILED DESCRIPTION:
The study will compare the efficacy of BWL + ER and BWL. Investigators will provide 6 months of treatment (BWL + ER or BWL) and will follow participants at 12-months post-treatment (total time = 18 months). Investigators will recruit adolescents with overweight and obesity and their parents. Dyads will be assessed at 5 timepoints: baseline (2 visits), mid-treatment (1 visit), post-treatment (2 visits), 6-month follow-up (2 visits), and 12-month follow-up (2 visits). Assessments will include the following for the adolescent and parent: anthropometry, emotion regulation, emotional inhibition, emotional eating, and adolescent-parent relationship measures. This program of research has the potential to advance the standard of practice for adolescents who are overweight or obese by providing alternative interventions.

We are currently offering online treatment groups to accommodate the CDC health and safety guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent age 13-16 years
* BMI percentile 85%85%-99.9% (adolescent only)
* Ability to read English at a minimum 6th grade level (both adolescent and parent); and willing to participate in a 6-month treatment and all assessments (both adolescent and parent)

Exclusion Criteria:

1. Current enrollment in a weight management program (Child and Parent);
2. Medication that is specifically prescribed for weight loss (Child and Parent);
3. Medical or psychiatric condition that may interfere with treatment participation (Child and Parent);
4. Regular use of compensatory behavior for weight loss (e.g., purging) during the past six months (Child and Parent);
5. Current pregnancy or lactating (Child and Parent);
6. Change in psychotropic medication during the previous three months (Child and Parent).

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 332 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Adolescent weight loss as measured by BMI, BMIz | Change from baseline to month 3, 6, 12, and 18.
Emotion Regulation Skills as measured by Ecological Momentary Assessment using State Difficulties in Emotion Regulation and International Positive and Negative Affect Schedule- Short form | Change from baseline to month 3, 6, 12, and 18.
Emotional Eating as measured by Emotional Eating Scale for children (EES-C) | Change from baseline to month 3, 6, 12, and 18.

SECONDARY OUTCOMES:
Parent BMI as measured by height and weight | Change from baseline to month 3, 6, 12, and 18.
Parent emotion regulation measured by Difficulties in Emotion Regulation Scale (DERS) | Change from baseline to month 3, 6, 12, and 18.
Parent emotional eating as measured by Emotional Eating Scale (EES) | Change from baseline to month 3, 6, 12, and 18.
Parent-adolescent relationship as measured by using: Inventory of Parents and Peer Attachment and Parental bonding assessment | Change from baseline to month 3, 6, 12, and 18.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, Ph.D., Principal Investigator — UCSD
Locations (2):
- United States (2):
  - UCSD Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California
  - Ambulatory Research Center - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boutelle KN, Manzano MA, Pasquale EK, Bernard RS, Strong DR, Rhee KE, Eichen DM, Engel S, Miller A, Peterson CB. Design of the FRESH-teen study: A randomized controlled trial evaluating an adapted emotion regulation weight loss program for adolescents with overweight or obesity and their parent. Contemp Clin Trials. 2024 Oct;145:107640. doi: 10.1016/j.cct.2024.107640. Epub 2024 Jul 28. PMID 39079614